CLINICAL TRIAL: NCT03260569
Title: Respiratory Mechanics Following Brain Injury: The Role of Inhaled Nitric Oxide
Brief Title: Inhaled Nitric Oxide in Brain Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael Goodman, Instructor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017 Goodman
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury
Keywords: Mechanical ventilation; Inhaled nitric oxide
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Following initial non-invasive measurements, patients will be randomized to either an active treatment (inhaled nitric oxide at 30 parts per million) or placebo (nitrogen only). After two hours, measurements will be reassessed. If the patient remains on the mechanical ventilator at 72 hours post-admission, a third set of non-invasive measurements will be taken.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both nitric oxide and placebo nitrogen will be made available in unmarked cylinders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inhaled Nitric Oxide (Active Comparator): Inhaled nitric oxide at 20 parts per million, administered once during first 36 hours following admission
  Interventions: Drug: Inhaled Nitric Oxide
- Placebo (Placebo Comparator): Nitrogen only, administered once during first 36 hours following admission
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Patients randomized to this arm will receive inhaled nitric oxide 20 parts per million.
  Arms: Inhaled Nitric Oxide
Drug: Placebo — Nitrogen plus oxygen
  Arms: Placebo

SUMMARY:
This study will evaluate the changes in respiratory mechanics following traumatic brain injury and determine the effect of inhaled nitric oxide on gas exchange.

DETAILED DESCRIPTION:
Intubation and mechanical ventilation are common treatments in the care of patients with traumatic brain injury (TBI). Intubation allows for airway control and facilitates removal of respiratory secretions. Mechanical ventilation allows control of arterial carbon dioxide to aid in control of intracranial pressure. Recent evidence suggests that lung protective ventilation (tidal volumes of 6 ml/kg of predicted body weight and moderate positive end expiratory pressure) improves outcomes following brain injury and reduces brain-lung cross talk.

The treatment of respiratory failure in TBI must balance the need to improve lung function with the negative consequences of increased intrathoracic pressure on mean arterial pressure, intracranial pressure and venous return. Traditional treatment of increasing positive end expiratory (PEEP) and mean airway pressure then, represent competing interests. Methods for improving arterial oxygenation while avoiding negative hemodynamic effects are needed.

The impact of head injury on respiratory mechanics has been studied in just a few clinical investigations. (1-3) Of note, the earliest of these noted that the ventilation perfusion (V/Q) matching following TBI was not the result of lung collapse or parenchymal lung disease but secondary to alterations in perfusion. There are three possibilities for this finding:

1. redistribution in regional perfusion, which is partially mediated by the hypothalamus
2. pulmonary microembolism, leading to increased dead space
3. lung surfactant depletion due to excessive sympathetic stimulation and hyperventilation.

The introduction of inhaled pulmonary vasodilators such as inhaled nitric oxide or aerosolized epoprostenol offer an opportunity to improve oxygenation in patients with TBI without increasing airway pressures in the face of V/Q inequalities.

This study will evaluate the changes in respiratory mechanics following TBI and determine the effect of inhaled nitric oxide on gas exchange.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission with traumatic brain injury (penetrating or blunt)
* Requirement for mechanical ventilation
* Glasgow Coma Score > 3

Exclusion Criteria:

* Brain death
* Expected survival < 48 hours
* Air leak (bronchopleural fistula, tracheal injury)
* Current inspired oxygen concentration (FiO2) > 0.65
* Hemodynamic instability (systolic blood pressure < 100 mm Hg, cardiac arrhythmia)
* Uncontrolled intracranial pressure (> 20 mm Hg)
* Spinal cord injury with hypotension
* Severe acute respiratory distress syndrome (ARDS) (PaO2/FiO2 < 100)
* Chest abbreviated injury score (AIS) > 3
* First rib fracture
* Flail chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schumacker PT, Rhodes GR, Newell JC, Dutton RE, Shah DM, Scovill WA, Powers SR. Ventilation-perfusion imbalance after head trauma. Am Rev Respir Dis. 1979 Jan;119(1):33-43. doi: 10.1164/arrd.1979.119.1.33. PMID 420436
- [Background] Cooper KR, Boswell PA. Accurate measurement of functional residual capacity and oxygen consumption of patients on mechanical ventilation. Anaesth Intensive Care. 1983 May;11(2):151-7. doi: 10.1177/0310057X8301100212. PMID 6346942
- [Background] Koutsoukou A, Perraki H, Raftopoulou A, Koulouris N, Sotiropoulou C, Kotanidou A, Orfanos S, Roussos C. Respiratory mechanics in brain-damaged patients. Intensive Care Med. 2006 Dec;32(12):1947-54. doi: 10.1007/s00134-006-0406-0. Epub 2006 Oct 20. PMID 17053881
- [Background] Gruber A, Reinprecht A, Illievich UM, Fitzgerald R, Dietrich W, Czech T, Richling B. Extracerebral organ dysfunction and neurologic outcome after aneurysmal subarachnoid hemorrhage. Crit Care Med. 1999 Mar;27(3):505-14. doi: 10.1097/00003246-199903000-00026. PMID 10199529
- [Background] Holland MC, Mackersie RC, Morabito D, Campbell AR, Kivett VA, Patel R, Erickson VR, Pittet JF. The development of acute lung injury is associated with worse neurologic outcome in patients with severe traumatic brain injury. J Trauma. 2003 Jul;55(1):106-11. doi: 10.1097/01.TA.0000071620.27375.BE. PMID 12855888
- [Background] Pelosi P, Severgnini P, Chiaranda M. An integrated approach to prevent and treat respiratory failure in brain-injured patients. Curr Opin Crit Care. 2005 Feb;11(1):37-42. doi: 10.1097/00075198-200502000-00006. PMID 15659943
- [Background] Garry PS, Ezra M, Rowland MJ, Westbrook J, Pattinson KT. The role of the nitric oxide pathway in brain injury and its treatment--from bench to bedside. Exp Neurol. 2015 Jan;263:235-43. doi: 10.1016/j.expneurol.2014.10.017. Epub 2014 Oct 29. PMID 25447937
- [Background] Terpolilli NA, Kim SW, Thal SC, Kuebler WM, Plesnila N. Inhaled nitric oxide reduces secondary brain damage after traumatic brain injury in mice. J Cereb Blood Flow Metab. 2013 Feb;33(2):311-8. doi: 10.1038/jcbfm.2012.176. Epub 2012 Nov 28. PMID 23188422
- [Background] Papadimos TJ, Medhkour A, Yermal S. Successful use of inhaled nitric oxide to decrease intracranial pressure in a patient with severe traumatic brain injury complicated by acute respiratory distress syndrome: a role for an anti-inflammatory mechanism? Scand J Trauma Resusc Emerg Med. 2009 Feb 17;17:5. doi: 10.1186/1757-7241-17-5. PMID 19222848
- [Background] Papadimos TJ. The beneficial effects of inhaled nitric oxide in patients with severe traumatic brain injury complicated by acute respiratory distress syndrome: a hypothesis. J Trauma Manag Outcomes. 2008 Jan 14;2(1):1. doi: 10.1186/1752-2897-2-1. PMID 18272001
- [Background] Vavilala MS, Roberts JS, Moore AE, Newell DW, Lam AM. The influence of inhaled nitric oxide on cerebral blood flow and metabolism in a child with traumatic brain injury. Anesth Analg. 2001 Aug;93(2):351-3 , 3rd contents page. doi: 10.1097/00000539-200108000-00023. PMID 11473859
- [Background] Dellinger RP, Zimmerman JL, Taylor RW, Straube RC, Hauser DL, Criner GJ, Davis K Jr, Hyers TM, Papadakos P. Effects of inhaled nitric oxide in patients with acute respiratory distress syndrome: results of a randomized phase II trial. Inhaled Nitric Oxide in ARDS Study Group. Crit Care Med. 1998 Jan;26(1):15-23. doi: 10.1097/00003246-199801000-00011. PMID 9428538
- [Background] Lundin S, Mang H, Smithies M, Stenqvist O, Frostell C. Inhalation of nitric oxide in acute lung injury: results of a European multicentre study. The European Study Group of Inhaled Nitric Oxide. Intensive Care Med. 1999 Sep;25(9):911-9. doi: 10.1007/s001340050982. PMID 10501745

RESULTS

PARTICIPANT FLOW:
Groups:
- in Haled Nitric Oxide: received nitric oxide
- Placebo: did not receive iNO
Period: Overall Study
Arm/Group | in Haled Nitric Oxide | Placebo
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inhaled Nitric Oxide: received nitric oxide
- Total: Total of all reporting groups
Arm/Group | Inhaled Nitric Oxide | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (17) | 49 (20) | 53 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Midwest
  participants
    United States | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: PaO2
Description: The primary endpoint is the difference in PO2
Time Frame: at Day 3 of the study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Inhaled Nitric Oxide | Placebo
Number analyzed (Participants) | 6 | 7
mmHg | 115 (10) | 95 (10)
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide vs Placebo; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Inhaled Nitric Oxide | Placebo
All-Cause Mortality (participants affected / at risk) | 3/6 | 2/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 0/6 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT03260569/Prot_SAP_003.pdf